CLINICAL TRIAL: NCT06557928
Title: Protocol for Evaluating Physiological and Psychological Adaptation Mechanisms in Tibetan Plateau Environments: A Clinical Study of Doctors From Peking Union Medical College Hospital
Brief Title: Protocol for Evaluating Physiological and Psychological Adaptation Mechanisms in Tibetan Plateau Environments
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Professor of Gastroenterology, Peking Union Medical College Hospital
Other Study IDs: 2022-I2M-1-003
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: High Altitude
Keywords: high altitude; adaptation; acclimatization
MeSH Terms: conditions — Altitude Sickness | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doctors to Tibet from Peking Union Medical College Hospital in 2024
  Interventions: Other: measurement
- Doctors to Tibet from Peking Union Medical College Hospital in 2025
  Interventions: Other: measurement

INTERVENTIONS:
Other: measurement — Measurement of multiple physiological indicators and psychological status and multi-omics study

SUMMARY:
This study is a single-center prospective observational study. It plans to use a series of physiological and medical instruments and international common physiological and psychological questionnaires. To dynamically detect the changes of physiological and psychological adaptability of doctors in Peking Union Medical College Hospital before leaving Beijing, 1-7 days after arriving at the plateau in Tibet during the acute phase of plateau hypoxic stress, 2 weeks, 3 months, 6 months, 12 months after staying in Tibet during the chronic phase of plateau hypoxic stress, and after returning to Beijing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 20-65 years
* They can sign a written informed consent and is willing to cooperate
* They have the qualification to aid Tibet and meet the basic requirements of physical examination for aid to Tibet

Exclusion Criteria:

* Age less than 20 years or more than 65 years
* Unable to sign a written informed consent or unwilling to cooperate
* They do not have the qualification for supporting Tibet or do not meet the basic requirements of medical examination for supporting Tibet

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Doctors in Tibet from Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
help understand the physiological mechanisms and psychological changes of hypoxic adaptation | 2024-5-27~2026-12-1
  This study is expected to increase our understanding of the physiological mechanisms and psychological changes of hypoxic adaptation mainly through analysis of multi-omics.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided